CLINICAL TRIAL: NCT03216902
Title: A Phase IIb, Randomized, Observer-Masked, Placebo- and Active-Controlled, Parallel-Group, Multinational and Multicenter Study Assessing the Safety and Efficacy of DE-126 Ophthalmic Solution in Subjects With Primary Open-Angle Glaucoma or Ocular Hypertension- Angel Study
Brief Title: A Phase IIb Safety and Efficacy Study of DE-126 Ophthalmic Solution in Primary Open-Angle Glaucoma or Ocular Hypertension- Angel Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Santen Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 012601IN
Record Dates: First submitted 2017-07-11; First posted 2017-07-13 (Actual); Results first posted 2020-10-23 (Actual); Last update posted 2020-10-23 (Actual); Status verified 2020-09

CONDITIONS: Open-angle Glaucoma, Ocular Hypertension
Keywords: Glaucoma
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension; Glaucoma | interventions — Latanoprost

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Placebo (Vehicle of DE-126) followed by high dose of DE-126 (Placebo Comparator)
  Interventions: Drug: Vehicle of DE-126 Ophthalmic Solution, high dose of DE-126 Ophthalmic Solution
- Ultra-low dose 0.0005% DE-126 (Experimental)
  Interventions: Drug: Topical ultra-low dose of DE-126 Ophthalmic Solution
- Low dose 0.001% DE-126 (Experimental)
  Interventions: Drug: Topical low dose of DE-126 Ophthalmic Solution
- Medium dose 0.002% DE-126 (Experimental)
  Interventions: Drug: Topical medium dose of DE-126 Ophthalmic Solution
- High dose 0.003% DE-126 (Experimental)
  Interventions: Drug: Topical high dose of DE-126 Ophthalmic Solution
- 0.005% Latanoprost (Active Comparator)
  Interventions: Drug: 0.005% Latanoprost Ophthalmic Solution

INTERVENTIONS:
Drug: Vehicle of DE-126 Ophthalmic Solution, high dose of DE-126 Ophthalmic Solution — Vehicle of DE-126 Ophthalmic Solution dosed once daily for 6weeks, followed by high dose of DE-126 dosed once daily for 6 additional weeks
  Arms: Placebo (Vehicle of DE-126) followed by high dose of DE-126
Drug: Topical ultra-low dose of DE-126 Ophthalmic Solution — Topical ultra-low dose of DE-126 Ophthalmic Solution dosed once daily for 12 weeks
  Arms: Ultra-low dose 0.0005% DE-126
Drug: Topical low dose of DE-126 Ophthalmic Solution — Topical low dose of DE-126 Ophthalmic Solution dosed once daily for 12 weeks
  Arms: Low dose 0.001% DE-126
Drug: Topical medium dose of DE-126 Ophthalmic Solution — Topical medium dose of DE-126 Ophthalmic Solution dosed once daily for 12 weeks
  Arms: Medium dose 0.002% DE-126
Drug: Topical high dose of DE-126 Ophthalmic Solution — Topical high dose of DE-126 Ophthalmic Solution dosed once daily for 12 weeks
  Arms: High dose 0.003% DE-126
Drug: 0.005% Latanoprost Ophthalmic Solution — 0.005% Latanoprost Ophthalmic Solution dosed once daily for 12 weeks
  Other Names: Xalatan®
  Arms: 0.005% Latanoprost

SUMMARY:
Treatment of elevated pressure in the eye (Intraocular pressure, or 'IOP') with eye drop medications has been shown to be effective in delaying or preventing the progression of glaucoma, and it is the only proven method for reducing the risk of glaucomatous visual field loss.

This study is being conducted to determine how well DE-126 ophthalmic solution works (efficacy) in safely lowering IOP when dosed as topical eyedrops. This study will evaluate the safety and efficacy of four (4) concentrations of DE-126, when compared with latanoprost (0.005%) eye drops in patients with primary open-angle glaucoma or ocular hypertension.

The IOP will be measured at 3 different times throughout the day, over 6 total visits during a 3-month treatment period (with up to 4 extra weeks observation if the patient must stop taking current eye drops to lower IOP). Safety assessments will be done throughout the study, including ocular signs and symptoms, vital signs, and clinical laboratory tests. While the most important time-point to measure IOP in this study and evaluate efficacy will be at the final study visit (month 3), IOP values will also be evaluated at other visits throughout the 3-month treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Provide signed written informed consent
* Diagnosis of POAG or OHT in both eyes
* Qualifying corrected visual acuity in each eye
* Qualifying central corneal thickness in each eye
* Qualifying Day 1 IOP measurement at 3 time-points in both eyes
* Qualifying Anterior chamber angle

Exclusion Criteria:

* History of ocular surgery specifically intended to lower IOP
* Subjects who cannot safely discontinue use of ocular hypotensive medications during the wait/washout period
* Advanced glaucoma in either eye
* Any corneal abnormality or other condition interfering with or preventing reliable Goldmann applanation tonometry
* Any ocular surgery or ocular laser treatment within 90 days prior to Visit 1 (Screening) and throughout the study in either eye
* Females who are pregnant, nursing, or planning a pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 241 (Actual)
Dates: Start 2017-07-25 (Actual); Primary Completion 2018-02-27 (Actual); Study Completion 2018-02-27 (Actual)

CONTACTS AND LOCATIONS:
Locations (17):
- United States (12):
  - Sall Research Medical Center, Inc, Artesia, California
  - North Valley Eye Medical Group, Mission Hills, California
  - Eye Research Foundation, INC, Newport Beach, California
  - North Bay Eye Associates, Inc., Petaluma, California
  - Shettle Eye Research, Inc., Largo, Florida
  - Clayton Eye Clinical Research, LLC, Morrow, Georgia
  - Coastal Research Associates, LLC, Roswell, Georgia
  - Rochester Ophthalmological Group, PC, Rochester, New York
  - Mundorf Eye Center, Charlotte, North Carolina
  - Cornerstone Health Care, LLC, High Point, North Carolina
  - Keystone Research Ltd SMO/Texan Eye, PA, Austin, Texas
  - Keystone Research LTD SMO/Medical Center Ophthalmology Assoc., San Antonio, Texas
- Japan (5):
  - Murakami Karindoh Hospital, Fukuoka-shi, Fukuoka
  - Nagasaka Eye Clinic, Nagoya-shi, Aichi
  - Sugiura Eye Clinic, Osaka-shi, Osaka
  - Sapporo Katoh Ophthalmology Clinic, Sapporo-shi, Hokkaido
  - Dogenzaka Kato Eye Clinic, Shibuya-ku, Tokyo

REFERENCES:
- [Derived] Wirta DL, Kuwayama Y, Lu F, Shao H, Odani-Kawabata N. Phase 2b, Randomized, 3-Month, Dose-Finding Study of Sepetaprost in Patients with Primary Open-Angle Glaucoma or Ocular Hypertension: The ANGEL Study. J Ocul Pharmacol Ther. 2022 Apr;38(3):240-251. doi: 10.1089/jop.2021.0077. Epub 2022 Feb 15. PMID 35167779

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo (Vehicle of DE-126) Followed by High Dose of DE-126 | 0.005% Latanoprost | Ultra-low Dose 0.0005% DE-126 | Low Dose 0.001% DE-126 | Medium Dose 0.002% DE-126 | High Dose 0.003% DE-126
Started | 22 | 44 | 43 | 43 | 44 | 45
Completed | 20 | 43 | 42 | 43 | 43 | 42
Not Completed | 2 | 1 | 1 | 0 | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo (Vehicle of DE-126) Followed by High Dose of DE-126 | 0.005% Latanoprost | Ultra-low Dose 0.0005% DE-126 | Low Dose 0.001% DE-126 | Medium Dose 0.002% DE-126 | High Dose 0.003% DE-126 | Total
Number analyzed (Participants) | 22 | 44 | 43 | 43 | 44 | 45 | 241
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.2 (11.24) | 64.4 (9.8) | 65.5 (13.30) | 63.7 (9.41) | 61.0 (11.84) | 63.8 (11.84) | 63.6 (11.22)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 24 | 26 | 22 | 25 | 25 | 135
  Male | 9 | 20 | 17 | 21 | 19 | 20 | 106
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 5 | 7 | 7 | 5 | 6 | 32
  Not Hispanic or Latino | 20 | 39 | 36 | 36 | 39 | 39 | 209
Region of Enrollment [Number; unit: participants]
  Japan | 11 | 21 | 20 | 20 | 21 | 21 | 114
  United States | 11 | 23 | 23 | 23 | 23 | 24 | 127

OUTCOME MEASURES:

1. Primary Outcome: Intraocular Pressure in the Study Eye at Month 3
Description: Intraocular Pressure (IOP),the fluid pressure inside the eye was measured by the Goldmann applanation tonometer in millimeters mercury (mmHg) at 3 time-points throughout the day.
Time Frame: 9:00, 13:00 and 17:00 at Month 3
Population: The number of participants is reduced due to missing data.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Placebo (Vehicle of DE-126) Followed by High Dose of DE-126 | 0.005% Latanoprost | Ultra-low Dose 0.0005% DE-126 | Low Dose 0.001% DE-126 | Medium Dose 0.002% DE-126 | High Dose 0.003% DE-126
Number analyzed (Participants) | 22 | 44 | 43 | 43 | 44 | 45
mmHg
  9:00: number analyzed (Participants) | 20 | 43 | 42 | 43 | 44 | 42
  9:00 | 18.8 (4.11) | 18.1 (3.73) | 19.7 (3.27) | 19.2 (3.37) | 17.6 (3.13) | 19.3 (2.92)
  13:00: number analyzed (Participants) | 20 | 43 | 42 | 43 | 44 | 42
  13:00 | 17.6 (3.18) | 17.3 (3.01) | 18.5 (2.98) | 18.1 (2.99) | 17.4 (2.39) | 18.7 (3.17)
  17:00: number analyzed (Participants) | 20 | 43 | 42 | 43 | 44 | 42
  17:00 | 17.8 (2.87) | 17.2 (3.10) | 18.3 (2.55) | 17.8 (2.93) | 16.7 (2.74) | 17.9 (2.82)

2. Secondary Outcome: Intraocular Pressure in the Study Eye at Week 6
Description: as for outcome 1
Time Frame: 9:00, 13:00 and 17:00 at Week 6
Population: The number of participants is reduced due to missing data. This endpoint is to test if one of four concentrations of DE-126 is superior to the placebo in lowering IOP at each specified timepoint (9:00, 13:00 and 17:00) at Week 6 compared to baseline. Therefore, 0.005% Latanoprost group is not included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Placebo (Vehicle of DE-126) Followed by High Dose of DE-126 | Ultra-low Dose 0.0005% DE-126 | Low Dose 0.001% DE-126 | Medium Dose 0.002% DE-126 | High Dose 0.003% DE-126
Number analyzed (Participants) | 22 | 43 | 43 | 44 | 45
mmHg
  9:00: number analyzed (Participants) | 20 | 42 | 43 | 44 | 44
  9:00 | 23.2 (0.66) | 19.0 (0.46) | 18.5 (0.46) | 18.7 (0.45) | 18.7 (0.45)
  13:00: number analyzed (Participants) | 20 | 42 | 43 | 44 | 44
  13:00 | 22.2 (0.61) | 18.2 (0.42) | 17.9 (0.42) | 17.3 (0.42) | 17.5 (0.41)
  17:00: number analyzed (Participants) | 20 | 42 | 43 | 44 | 44
  17:00 | 21.6 (0.62) | 17.8 (0.43) | 17.9 (0.43) | 16.6 (0.42) | 17.4 (0.42)
Statistical Analysis 1: Comparison: Placebo (Vehicle of DE-126) Followed by High Dose of DE-126 vs Ultra-low Dose 0.0005% DE-126; This endpoint is to test if one of four concentrations of DE-126 is superior to the placebo in lowering IOP at each specified timepoint (9:00, 13:00 and 17:00) at Week 6 compared to baseline. Therefore, 0.005% Latanoprost group is not included in the analysis; Test type: Superiority — Claim superiority of DE-126 compare to Placebo at 3 timepoints (9:00, 13:00 and 17:00); p < 0.0001, t-test, 2 sided — P value is adjusted for multiple comparisons using Hochberg step-up procedure
Statistical Analysis 2: Comparison: Placebo (Vehicle of DE-126) Followed by High Dose of DE-126 vs Low Dose 0.001% DE-126; [analysis description as in outcome 2, analysis 1]; Test type: Superiority — Claim superiority of DE-126 compare to Placebo at 3 timepoints (9:00, 13:00 and 17:00); p < 0.0001, t-test, 2 sided — P value is adjusted for multiple comparisons using Hochberg step-up procedure
Statistical Analysis 3: Comparison: Placebo (Vehicle of DE-126) Followed by High Dose of DE-126 vs Medium Dose 0.002% DE-126; [analysis description as in outcome 2, analysis 1]; Test type: Superiority — Claim superiority of DE-126 compare to Placebo at 3 timepoints (9:00, 13:00 and 17:00); p < 0.0001, t-test, 2 sided — P value is adjusted for multiple comparisons using Hochberg step-up procedure
Statistical Analysis 4: Comparison: Placebo (Vehicle of DE-126) Followed by High Dose of DE-126 vs High Dose 0.003% DE-126; [analysis description as in outcome 2, analysis 1]; Test type: Superiority — Claim superiority of DE-126 compare to Placebo at 3 timepoints (9:00, 13:00 and 17:00); p < 0.0001, t-test, 2 sided — P value is adjusted for multiple comparisons using Hochberg step-up procedure

3. Secondary Outcome: Intraocular Pressure in the Study Eye at Week 1 and Week 2
Description: as for outcome 1
Time Frame: 9:00, 13:00 and 17:00 at Week 1 and Week 2
Population: The number of participants is reduced due to missing data.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Placebo (Vehicle of DE-126) Followed by High Dose of DE-126 | 0.005% Latanoprost | Ultra-low Dose 0.0005% DE-126 | Low Dose 0.001% DE-126 | Medium Dose 0.002% DE-126 | High Dose 0.003% DE-126
Number analyzed (Participants) | 22 | 44 | 43 | 43 | 44 | 45
mmHg
  Week1 9:00: number analyzed (Participants) | 22 | 44 | 42 | 43 | 44 | 45
  Week1 9:00 | 22.8 (3.99) | 17.7 (2.67) | 19.4 (3.32) | 18.9 (2.82) | 18.1 (2.99) | 18.0 (2.66)
  Week1 13:00: number analyzed (Participants) | 22 | 44 | 42 | 43 | 43 | 45
  Week1 13:00 | 22.8 (3.66) | 17.5 (2.25) | 18.7 (3.28) | 18.6 (3.29) | 17.1 (2.65) | 17.6 (3.08)
  Week1 17:00: number analyzed (Participants) | 22 | 44 | 42 | 43 | 43 | 44
  Week1 17:00 | 21.6 (3.94) | 17.4 (2.43) | 18.1 (2.94) | 18.5 (3.23) | 16.9 (2.96) | 17.2 (2.53)
  Week 2 9:00: number analyzed (Participants) | 21 | 44 | 43 | 43 | 44 | 44
  Week 2 9:00 | 22.7 (3.70) | 17.6 (3.33) | 19.4 (3.62) | 18.7 (2.73) | 17.9 (3.11) | 18.3 (3.13)
  Week 2 13:00: number analyzed (Participants) | 21 | 44 | 43 | 43 | 44 | 44
  Week 2 13:00 | 22.0 (3.13) | 17.4 (2.45) | 18.2 (2.93) | 18.1 (2.77) | 17.2 (2.57) | 17.6 (2.80)
  Week2 17:00: number analyzed (Participants) | 21 | 44 | 43 | 43 | 44 | 44
  Week2 17:00 | 21.9 (3.93) | 16.9 (2.49) | 18.2 (2.94) | 17.8 (2.33) | 16.7 (2.89) | 17.3 (2.59)

4. Secondary Outcome: Mean Diurnal Intraocular Pressure in the Study Eye at Each Post-baseline Visit
Description: Mean Diurnal IOP was defined as the mean of the IOP values at the three schedules timepoints (9:00, 13:00 and 17:00) at that visit for that subject.
Time Frame: Week 1, Week 2, Week 6 and Month 3.
Population: The number of participants is reduced due to missing data.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Placebo (Vehicle of DE-126) Followed by High Dose of DE-126 | 0.005% Latanoprost | Ultra-low Dose 0.0005% DE-126 | Low Dose 0.001% DE-126 | Medium Dose 0.002% DE-126 | High Dose 0.003% DE-126
Number analyzed (Participants) | 22 | 44 | 43 | 43 | 44 | 45
mmHg
  Week 1: number analyzed (Participants) | 22 | 44 | 42 | 43 | 43 | 44
  Week 1 | 22.4 (3.48) | 17.5 (2.12) | 18.8 (2.95) | 18.7 (2.88) | 17.4 (2.64) | 17.6 (2.59)
  Week 2: number analyzed (Participants) | 21 | 44 | 43 | 43 | 44 | 44
  Week 2 | 22.2 (3.33) | 17.3 (2.51) | 18.6 (2.92) | 18.2 (2.37) | 17.3 (2.58) | 17.7 (2.52)
  Week 6: number analyzed (Participants) | 20 | 43 | 42 | 43 | 44 | 44
  Week 6 | 21.7 (2.90) | 17.3 (2.80) | 18.4 (2.40) | 18.1 (2.50) | 17.5 (2.69) | 17.8 (2.69)
  Month 3: number analyzed (Participants) | 20 | 43 | 42 | 43 | 44 | 42
  Month 3 | 18.1 (3.14) | 17.5 (2.98) | 18.8 (2.66) | 18.4 (2.94) | 17.2 (2.47) | 18.6 (2.71)

5. Secondary Outcome: Change From Baseline (CFB) in Mean Diurnal Intraocular Pressure in the Study Eye at Each Post-baseline Visit
Description: as for outcome 4
Time Frame: Week 1, Week 2, Week 6 and Month 3.
Population: The number of participants is reduced due to missing data.
Measure: Mean (Standard Deviation); unit: mmHg
Groups:
- 0.001% Low Dose DE-126: Topical low dose of DE-126 Ophthalmic Solution: Topical low dose of DE-126 Ophthalmic Solution dosed once daily for 12 weeks
Arm/Group | Placebo (Vehicle of DE-126) Followed by High Dose of DE-126 | 0.005% Latanoprost | Ultra-low Dose 0.0005% DE-126 | 0.001% Low Dose DE-126 | Medium Dose 0.002% DE-126 | High Dose 0.003% DE-126
Number analyzed (Participants) | 22 | 44 | 43 | 43 | 44 | 45
mmHg
  Week 1: number analyzed (Participants) | 22 | 44 | 42 | 43 | 43 | 44
  Week 1 | -2.1 (2.13) | -6.7 (2.98) | -5.5 (2.41) | -5.6 (2.84) | -6.7 (3.19) | -6.6 (2.92)
  Week 2: number analyzed (Participants) | 21 | 44 | 43 | 43 | 44 | 44
  Week 2 | -2.0 (2.15) | -7.0 (3.13) | -5.8 (3.02) | -6.0 (2.35) | -6.9 (2.87) | -6.5 (2.94)
  Week 6: number analyzed (Participants) | 20 | 43 | 42 | 43 | 44 | 44
  Week 6 | -2.3 (2.49) | -7.0 (3.09) | -5.9 (2.73) | -6.1 (2.59) | -6.6 (3.08) | -6.4 (2.68)
  Month 3: number analyzed (Participants) | 20 | 43 | 42 | 43 | 44 | 42
  Month 3 | -5.9 (2.65) | -6.7 (3.24) | -5.5 (2.11) | -5.9 (2.71) | -6.9 (2.96) | -5.5 (2.67)

6. Secondary Outcome: Percent Change From Baseline (CFB) in Mean Diurnal Intraocular Pressure in the Study Eye at Each Post-baseline Visit
Description: as for outcome 4
Time Frame: Week 1, Week 2, Week 6 and Month 3.
Population: The number of participants is reduced due to missing data.
Measure: Mean (Standard Deviation); unit: Percentage of change
Arm/Group | Placebo (Vehicle of DE-126) Followed by High Dose of DE-126 | 0.005% Latanoprost | Ultra-low Dose 0.0005% DE-126 | Low Dose 0.001% DE-126 | Medium Dose 0.002% DE-126 | High Dose 0.003% DE-126
Number analyzed (Participants) | 22 | 44 | 43 | 43 | 44 | 45
Percentage of change
  Week 1: number analyzed (Participants) | 22 | 44 | 42 | 43 | 43 | 44
  Week 1 | -8.6 (8.15) | -27.3 (10.60) | -22.8 (9.59) | -22.9 (10.78) | -27.4 (11.48) | -27.0 (11.12)
  Week 2: number analyzed (Participants) | 21 | 44 | 43 | 43 | 44 | 44
  Week 2 | -8.6 (8.74) | -28.3 (11.05) | -23.5 (11.28) | -24.7 (8.90) | -28.2 (10.48) | -26.4 (11.27)
  Week 6: number analyzed (Participants) | 20 | 43 | 42 | 43 | 44 | 44
  Week 6 | -9.4 (10.31) | -28.5 (11.23) | -24.0 (9.58) | -25.1 (9.83) | -27.2 (10.72) | -26.2 (10.51)
  Month 3: number analyzed (Participants) | 20 | 43 | 42 | 43 | 44 | 42
  Month 3 | -24.7 (11.26) | -27.5 (12.11) | -22.6 (8.22) | -24.1 (10.45) | -28.4 (10.54) | -22.7 (10.79)

7. Secondary Outcome: Change From Baseline (CFB) in Intraocular Pressure in the Study Eye at Three Time Points at Each Post-baseline Visit
Description: as for outcome 1
Time Frame: 9:00, 13:00 and 17:00 at Week 1, Week 2, Week 6 and Month 3.
Population: The number of participants is reduced due to missing data.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Placebo (Vehicle of DE-126) Followed by High Dose of DE-126 | 0.005% Latanoprost | Ultra-low Dose 0.0005% DE-126 | Low Dose 0.001% DE-126 | Medium Dose 0.002% DE-126 | High Dose 0.003% DE-126
Number analyzed (Participants) | 22 | 44 | 43 | 43 | 44 | 45
mmHg
  Week 1 9:00: number analyzed (Participants) | 22 | 44 | 42 | 43 | 44 | 45
  Week 1 9:00 | -2.1 (2.68) | -7.3 (3.65) | -5.3 (2.65) | -6.0 (3.10) | -6.7 (3.70) | -6.6 (3.24)
  Week 1 13:00: number analyzed (Participants) | 22 | 44 | 42 | 43 | 43 | 45
  Week 1 13:00 | -1.2 (2.73) | -6.8 (3.35) | -5.7 (2.73) | -5.6 (3.26) | -6.8 (3.59) | -6.7 (3.63)
  Week 1 17:00: number analyzed (Participants) | 22 | 44 | 42 | 43 | 43 | 44
  Week 1 17:00 | -2.8 (2.81) | -6.2 (3.33) | -5.6 (2.83) | -5.2 (3.62) | -6.7 (3.60) | -6.4 (2.98)
  Week 2 9:00: number analyzed (Participants) | 21 | 44 | 43 | 43 | 44 | 44
  Week 2 9:00 | -1.9 (2.66) | -7.4 (4.03) | -5.5 (3.52) | -6.2 (3.00) | -6.9 (3.32) | -6.4 (3.66)
  Week 2 13:00: number analyzed (Participants) | 21 | 44 | 43 | 43 | 44 | 44
  Week 2 13:00 | -1.8 (2.89) | -6.8 (3.02) | -6.2 (3.36) | -6.0 (2.62) | -6.8 (3.27) | -6.7 (3.22)
  Week 2 17:00: number analyzed (Participants) | 21 | 44 | 43 | 43 | 44 | 44
  Week 2 17:00 | -2.4 (2.57) | -6.7 (3.39) | -5.7 (3.36) | -5.8 (2.52) | -6.9 (3.29) | -6.3 (3.15)
  Week 6 9:00: number analyzed (Participants) | 20 | 44 | 42 | 43 | 44 | 44
  Week 6 9:00 | -2.0 (2.59) | -7.0 (3.84) | -5.7 (3.03) | -6.4 (2.83) | -6.1 (3.21) | -6.1 (3.55)
  Week 6 13:00: number analyzed (Participants) | 20 | 43 | 42 | 43 | 44 | 44
  Week 6 13:00 | -2.1 (2.66) | -7.0 (3.30) | -6.1 (3.65) | -6.2 (2.64) | -6.8 (3.67) | -6.8 (3.11)
  Week 6 17:00: number analyzed (Participants) | 20 | 43 | 42 | 43 | 44 | 44
  Week 6 17:00 | -2.7 (3.33) | -6.8 (3.38) | -5.9 (2.56) | -5.7 (3.30) | -7.0 (3.36) | -6.2 (3.16)
  Month 3 at 9:00: number analyzed (Participants) | 20 | 43 | 42 | 43 | 44 | 42
  Month 3 at 9:00 | -5.6 (3.21) | -6.9 (3.84) | -5.1 (2.42) | -5.7 (3.08) | -7.2 (3.32) | -5.4 (3.41)
  Month 3 at 13:00: number analyzed (Participants) | 20 | 43 | 42 | 43 | 44 | 42
  Month 3 at 13:00 | -6.0 (3.28) | -6.9 (3.25) | -5.9 (2.49) | -6.0 (2.97) | -6.7 (3.34) | -5.5 (3.53)
  Month 3 at 17:00: number analyzed (Participants) | 20 | 43 | 42 | 43 | 44 | 42
  Month 3 at 17:00 | -6.1 (2.74) | -6.4 (3.63) | -5.4 (2.74) | -5.8 (3.12) | -6.9 (3.48) | -5.5 (2.93)

8. Secondary Outcome: Percent Change From Baseline (CFB) in Intraocular Pressure in the Study Eye at Three Time Points at Each Post-baseline Visit
Description: as for outcome 1
Time Frame: 9:00, 13:00 and 17:00 at Week 1, Week 2, Week 6 and Month 3.
Population: The number of participants is reduced due to missing data.
Measure: Mean (Standard Deviation); unit: Percentage of change in IOP
Arm/Group | Placebo (Vehicle of DE-126) Followed by High Dose of DE-126 | 0.005% Latanoprost | Ultra-low Dose 0.0005% DE-126 | Low Dose 0.001% DE-126 | Medium Dose 0.002% DE-126 | High Dose 0.003% DE-126
Number analyzed (Participants) | 22 | 44 | 43 | 43 | 44 | 45
Percentage of change in IOP
  Week 1 9:00: number analyzed (Participants) | 22 | 44 | 42 | 43 | 44 | 45
  Week 1 9:00 | -8.7 (9.58) | -28.5 (12.00) | -21.6 (10.44) | -23.7 (11.01) | -26.5 (12.64) | -26.5 (11.41)
  Week 1 13:00: number analyzed (Participants) | 22 | 44 | 42 | 43 | 43 | 45
  Week 1 13:00 | -5.3 (10.75) | -27.3 (11.41) | -23.3 (11.09) | -22.8 (12.54) | -28.0 (12.43) | -27.0 (13.50)
  Week 1 17:00: number analyzed (Participants) | 22 | 44 | 42 | 43 | 43 | 44
  Week 1 17:00 | -11.5 (10.56) | -25.7 (12.62) | -23.4 (10.96) | -21.5 (14.33) | -27.9 (13.10) | -26.8 (11.24)
  Week 2 9:00: number analyzed (Participants) | 21 | 44 | 43 | 43 | 44 | 44
  Week 2 9:00 | -7.8 (10.30) | -28.9 (13.13) | -21.7 (13.84) | -24.5 (10.62) | -27.4 (11.69) | -25.6 (13.56)
  Week 2 13:00: number analyzed (Participants) | 21 | 44 | 43 | 43 | 44 | 44
  Week 2 13:00 | -7.5 (12.08) | -27.8 (10.89) | -25.1 (12.42) | -24.9 (10.09) | -27.8 (11.83) | -27.0 (11.93)
  Week 2 17:00: number analyzed (Participants) | 21 | 44 | 43 | 43 | 44 | 44
  Week 2 17:00 | -9.9 (10.16) | -27.8 (12.69) | -23.5 (12.42) | -24.4 (9.53) | -28.8 (12.48) | -26.3 (11.95)
  Week 6 9:00: number analyzed (Participants) | 20 | 44 | 42 | 43 | 44 | 44
  Week 6 9:00 | -8.4 (10.71) | -27.5 (12.44) | -22.8 (10.71) | -25.3 (9.93) | -24.4 (11.45) | -24.3 (13.78)
  Week 6 13:00: number analyzed (Participants) | 20 | 43 | 42 | 43 | 44 | 44
  Week 6 13:00 | -8.6 (10.89) | -28.8 (12.25) | -24.5 (12.69) | -25.6 (9.85) | -27.7 (12.16) | -27.8 (11.27)
  Week 6 17:00: number analyzed (Participants) | 20 | 43 | 42 | 43 | 44 | 44
  Week 6 17:00 | -11.1 (13.12) | -28.4 (12.62) | -24.6 (9.63) | -24.0 (12.84) | -29.4 (11.86) | -26.1 (12.12)
  Month 3 at 9:00: number analyzed (Participants) | 20 | 43 | 42 | 43 | 44 | 42
  Month 3 at 9:00 | -23.3 (13.33) | -27.3 (13.11) | -20.6 (9.64) | -22.8 (11.48) | -28.8 (11.66) | -21.4 (12.63)
  Month 3 at 13:00: number analyzed (Participants) | 20 | 43 | 42 | 43 | 44 | 42
  Month 3 at 13:00 | -25.3 (13.15) | -28.2 (12.30) | -24.2 (10.00) | -24.8 (11.33) | -27.3 (11.73) | -22.5 (13.24)
  Month 3 at 17:00: number analyzed (Participants) | 20 | 43 | 42 | 43 | 44 | 42
  Month 3 at 17:00 | -25.4 (11.12) | -26.8 (14.63) | -22.7 (10.37) | -24.3 (12.06) | -28.7 (12.82) | -23.4 (11.96)

9. Secondary Outcome: Percentage of Subjects With Mean Diurnal Intraocular Pressure Reduction From Baseline ≥ 20%, 25% and 30% in the Study Eye at Each Post-baseline Visit
Description: A Subject was a responder if the percent reduction from baseline in mean diurnal IOP in the study eye was ≥ 20%.
  A Subject was a responder if the percent reduction from baseline in mean diurnal IOP in the study eye was ≥ 25%.
  A Subject was a responder if the percent reduction from baseline in mean diurnal IOP in the study eye was ≥ 30%.
Time Frame: WeeK 1, Week 2, Week 6 and Month 3.
Population: The number of participants is reduced due to missing data.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (Vehicle of DE-126) Followed by High Dose of DE-126 | 0.005% Latanoprost | Ultra-low Dose 0.0005% DE-126 | Low Dose 0.001% DE-126 | Medium Dose 0.002% DE-126 | High Dose 0.003% DE-126
Number analyzed (Participants) | 22 | 44 | 42 | 43 | 44 | 45
Participants
  Week 1- At Least 20% Reduction: number analyzed (Participants) | 22 | 44 | 42 | 43 | 44 | 44
  Week 1- At Least 20% Reduction | 2 | 36 | 22 | 28 | 31 | 34
  Week 1- At Least 25% Reduction: number analyzed (Participants) | 22 | 44 | 42 | 43 | 44 | 44
  Week 1- At Least 25% Reduction | 0 | 23 | 18 | 15 | 25 | 27
  Week 1- At Least 30% Reduction: number analyzed (Participants) | 22 | 44 | 42 | 43 | 44 | 44
  Week 1- At Least 30% Reduction | 0 | 16 | 9 | 8 | 14 | 18
  Week 2- At Least 20% Reduction: number analyzed (Participants) | 21 | 44 | 42 | 43 | 44 | 44
  Week 2- At Least 20% Reduction | 0 | 38 | 27 | 26 | 31 | 33
  Week 2- At Least 25% Reduction: number analyzed (Participants) | 21 | 44 | 42 | 43 | 44 | 44
  Week 2- At Least 25% Reduction | 0 | 27 | 21 | 22 | 27 | 24
  Week 2- At Least 30% Reduction: number analyzed (Participants) | 21 | 44 | 42 | 43 | 44 | 44
  Week 2- At Least 30% Reduction | 0 | 20 | 13 | 13 | 17 | 15
  Week 6- At Least 20% Reduction: number analyzed (Participants) | 20 | 43 | 42 | 43 | 44 | 44
  Week 6- At Least 20% Reduction | 3 | 37 | 30 | 28 | 30 | 28
  Week 6- At Least 25% Reduction: number analyzed (Participants) | 20 | 43 | 42 | 43 | 44 | 44
  Week 6- At Least 25% Reduction | 1 | 26 | 17 | 22 | 22 | 26
  Week 6- At Least 30% Reduction: number analyzed (Participants) | 20 | 43 | 42 | 43 | 44 | 44
  Week 6- At Least 30% Reduction | 1 | 19 | 12 | 18 | 15 | 14
  Month 3- At Least 20% Reduction: number analyzed (Participants) | 0 | 43 | 42 | 43 | 44 | 42
  Month 3- At Least 20% Reduction |  | 36 | 28 | 27 | 37 | 23
  Month 3- At Least 25% Reduction: number analyzed (Participants) | 0 | 43 | 42 | 43 | 44 | 42
  Month 3- At Least 25% Reduction |  | 23 | 15 | 22 | 28 | 18
  Month 3- At Least 30% Reduction: number analyzed (Participants) | 0 | 43 | 42 | 43 | 44 | 42
  Month 3- At Least 30% Reduction |  | 16 | 7 | 11 | 16 | 10

10. Secondary Outcome: Percentage of Subjects With Mean Diurnal Intraocular Pressure ≤ 18 mmHg in the Study Eye at Each Post-baseline Visit
Description: A subject was a responder if the mean diurnal IOP in the study eye was ≤ 18 mmHg.
Time Frame: Week 1, Week 2, Week 6 and Month 3.
Population: The number of participants is reduced due to missing data.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (Vehicle of DE-126) Followed by High Dose of DE-126 | 0.005% Latanoprost | Ultra-low Dose 0.0005% DE-126 | Low Dose 0.001% DE-126 | Medium Dose 0.002% DE-126 | High Dose 0.003% DE-126
Number analyzed (Participants) | 22 | 44 | 43 | 43 | 44 | 45
Participants
  Week 1 -Reduced to 18 mmHg or Lower: number analyzed (Participants) | 22 | 44 | 42 | 43 | 43 | 44
  Week 1 -Reduced to 18 mmHg or Lower | 0 | 29 | 16 | 20 | 26 | 30
  Week 2 -Reduced to 18 mmHg or Lower: number analyzed (Participants) | 21 | 44 | 43 | 43 | 44 | 44
  Week 2 -Reduced to 18 mmHg or Lower | 1 | 30 | 18 | 22 | 27 | 23
  Week 6 -Reduced to 18 mmHg or Lower: number analyzed (Participants) | 20 | 43 | 42 | 43 | 44 | 44
  Week 6 -Reduced to 18 mmHg or Lower | 2 | 27 | 24 | 22 | 25 | 23
  Month 3 -Reduced to 18 mmHg or Lower: number analyzed (Participants) | 0 | 43 | 42 | 43 | 44 | 42
  Month 3 -Reduced to 18 mmHg or Lower |  | 30 | 18 | 19 | 27 | 14

ADVERSE EVENTS:
Time Frame: Reporting time frame is from Inform Consent to end of the study at Month3.
Groups:
- Placebo P1: Vehicle of DE-126 Ophthalmic Solution, high dose of DE-126 Ophthalmic Solution: Vehicle of DE-126 Ophthalmic Solution dosed once daily for 6weeks.
- Placebo P2: Vehicle of DE-126 Ophthalmic Solution, high dose of DE-126 Ophthalmic Solution: Vehicle of DE-126 Ophthalmic Solution treatment arm dosed by high dose of DE-126 dosed once daily from w6 to month3.
- Ultra-low Dose DE-126: Topical ultra-low dose of DE-126 Ophthalmic Solution: Topical ultra-low dose of DE-126 Ophthalmic Solution dosed once daily for 12 weeks
- Low Dose DE-126: Topical low dose of DE-126 Ophthalmic Solution: Topical low dose of DE-126 Ophthalmic Solution dosed once daily for 12 weeks
- Medium Dose DE-126: Topical medium dose of DE-126 Ophthalmic Solution: Topical medium dose of DE-126 Ophthalmic Solution dosed once daily for 12 weeks
- High Dose of DE-126: Topical high dose of DE-126 Ophthalmic Solution: Topical high dose of DE-126 Ophthalmic Solution dosed once daily for 12 weeks
- High Dose of DE-126 Total: Summarizes columns High dose of DE-126 and Placebo P2
- DE-126 Total: Total summarizes columns Ultra Low Dose, Low Dose, Medium Dose, High Dose and Placebo P2.
Arm/Group | Placebo P1 | Placebo P2 | 0.005% Latanoprost | Ultra-low Dose DE-126 | Low Dose DE-126 | Medium Dose DE-126 | High Dose of DE-126 | High Dose of DE-126 Total | DE-126 Total
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/20 | 0/44 | 0/43 | 0/43 | 0/44 | 0/45 | 0/65 | 0/195
Serious Adverse Events (participants affected / at risk) | 1/22 | 0/20 | 0/44 | 0/43 | 0/43 | 0/44 | 0/45 | 0/65 | 0/195
Other Adverse Events (participants affected / at risk) | 2/22 | 10/20 | 18/44 | 13/43 | 12/43 | 10/44 | 12/45 | 22/65 | 57/195
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo P1 (N=22) | Placebo P2 (N=20) | 0.005% Latanoprost (N=44) | Ultra-low Dose DE-126 (N=43) | Low Dose DE-126 (N=43) | Medium Dose DE-126 (N=44) | High Dose of DE-126 (N=45) | High Dose of DE-126 Total (N=65) | DE-126 Total (N=195)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo P1 (N=22) | Placebo P2 (N=20) | 0.005% Latanoprost (N=44) | Ultra-low Dose DE-126 (N=43) | Low Dose DE-126 (N=43) | Medium Dose DE-126 (N=44) | High Dose of DE-126 (N=45) | High Dose of DE-126 Total (N=65) | DE-126 Total (N=195)
Cataract (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 2 (2)
Conjunctival Hyperaemia (Eye disorders) | 0 (0) | 2 (2) | 12 (13) | 5 (8) | 5 (5) | 9 (10) | 7 (8) | 9 (10) | 28 (33)
Eye Irritation (Eye disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 3 (4)
Eye Pruritus (Eye disorders) | 0 (0) | 0 (0) | 5 (5) | 2 (2) | 1 (1) | 0 (0) | 5 (5) | 5 (5) | 8 (8)
Growth Of Eyelashes (Eye disorders) | 0 (0) | 1 (1) | 2 (2) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 6 (6)
Lacrimation Increased (Eye disorders) | 0 (0) | 1 (1) | 3 (4) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 3 (4)
Instillation Site Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 1 (1) | 1 (1) | 5 (5)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Alveolar Osteitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 3 (3)
Upper Respiratory Tract Infection (Infections and infestations) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 2 (2) | 5 (5)
Viral Upper Respiratory Tract Infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 3 (3) | 2 (2) | 1 (1) | 2 (2) | 2 (2) | 8 (8)
Hepatic Enzyme Increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hypertonic Bladder (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Skin Lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Phlebitis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If Institution/Principal Investigator wishes to publish findings, they must submit draft to Santen at least 30 days prior, deleting Confidential Information if requested. Santen must be allowed up to ninety (90) days to determine if patent application is to be filed. Santen has right to first publication of Multi-Center Research results, but if publication doesn't occur within 12 months after completion, Institution/Principal Investigator may individually publish site's results.

DOCUMENTS (2):
  • Study Protocol (2017-06-16): https://cdn.clinicaltrials.gov/large-docs/02/NCT03216902/Prot_000.pdf
  • Statistical Analysis Plan (2018-03-27): https://cdn.clinicaltrials.gov/large-docs/02/NCT03216902/SAP_001.pdf